CLINICAL TRIAL: NCT02921360
Title: Randomised Controlled Prospective Trial of Early Administration of Aspirin After Systemic Thrombolysis in Acute Ischemic Stroke
Brief Title: Early Administration of Aspirin in Patients With Acute Ischemic Stroke Treated With Systemic Thrombolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: City Clinical Hospital No. 67, Moscow, Russia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GKB67-001
Record Dates: First submitted 2016-09-12; First posted 2016-10-03 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Stroke; Brain Ischemia
Keywords: thrombolytic therapy; tissue plasminogen activator; aspirin
MeSH Terms: conditions — Stroke; Brain Ischemia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- 12 hours (Experimental): Non-contrast CT and CT-angiography are performed in 11 hours after thrombolysis. In case no haematoma is found, patient would receive 100 mg of acetylsalicylic acid per os daily starting from 12 hours after thrombolysis
  Interventions: Drug: acetylsalicylic acid
- 24 hours (No Intervention): Non-contrast CT and CT-angiography are performed in 23 hours after thrombolysis. In case no haematoma is found, patient would receive 100 mg of acetylsalicylic acid per os daily starting from 24 hours after thrombolysis

INTERVENTIONS:
Drug: acetylsalicylic acid
  Other Names: aspirin
  Arms: 12 hours

SUMMARY:
The aim of this study is to determine whether early administration of aspirin in acute ischemic stroke patients treated with systemic thrombolysis is safe and can improve outcomes due to decreasing the number of early rethromboses.

DETAILED DESCRIPTION:
According to the current guidelines (European Stroke Organisation, 2009; American Heart Association-American Stroke Association, 2013) on the systemic thrombolysis in ischemic stroke patients it is recommended (class C) to start antithrombotic therapy (including antiplatelets and anticoagulants) when 24 hours go after alteplase (rtPA, recombinant tissue plasminogen activator) administration. Meanwhile rtPA has wery short lifetime in blood (T1/2 4-6 minutes). Some retrospective studies have found that early administration of antithrombotics (8-16 hours) after systemic thrombolysis can improve functional outcome and does not increase the risk of haemorrhage.

The investigators suggest a controlled prospective trial to recognise risks and benefits of early administration of aspirin (in 12 hours) after rtPA therapy in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke patients treated with rtPA
* mRS score before current stroke <4
* NIHSS score after rtPA treatment <25

Exclusion Criteria:

* contraindications for treatment with aspirin
* contraindications fot iodinated radiocontrast agents administration
* intracranial haemorrhage after rtPA treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 3 month
ischemic events | 3 month
  acute myocardial infarction and ischemic stroke
haemorrhagic events | 7 days
  intracerebral haemorrhage, gastrointestinal bleeding, other significant haemorrhage

SECONDARY OUTCOMES:
functional outcome | 3 month
  defined by modified Rankin scale
artery reocclusion | 7 days
  verified by CT-angiography

REFERENCES:
- [Background] Amaro S, Llull L, Urra X, Obach V, Cervera A, Chamorro A. Risks and benefits of early antithrombotic therapy after thrombolytic treatment in patients with acute stroke. PLoS One. 2013 Aug 8;8(8):e71132. doi: 10.1371/journal.pone.0071132. eCollection 2013. PMID 23951093